CLINICAL TRIAL: NCT01696045
Title: Phase 2 Study of Ipilimumab in Children and Adolescents (12 to < 18 Years) With Previously Treated or Untreated, Unresectable Stage III or Stage IV Malignant Melanoma
Brief Title: Phase 2 Study of Ipilimumab in Children and Adolescents (12 to < 18 Years) With Previously Treated or Untreated, Unresectable Stage III or Stage lV Malignant Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-178; 2012-002249-39 (EudraCT Number)
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-07

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ipilimumab 3 mg/kg (Experimental): Ipilimumab (3 mg/kg) was administered intravenously (IV) over 90 minutes on Day 1 of each 21-day cycle for 4 cycles.
  Interventions: Biological: Ipilimumab
- Ipilimumab 10 mg/kg (Experimental): Ipilimumab (10 mg/kg) was administered intravenously (IV) over 90 minutes on Day 1 of each 21-day cycle for 4 cycles.
  Interventions: Biological: Ipilimumab

INTERVENTIONS:
Biological: Ipilimumab
  Other Names: Yervoy; BMS- 734016

SUMMARY:
The purpose of the study is to comply with the Pediatric Investigation Plan requirements of Ipilimumab

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* 12 < 18 years of age
* Previously treated or untreated, unresectable Stage III or Stage IV malignant melanoma
* Karnofsky Performance Status (KPS) or Lansky Score ≥ 50

Exclusion Criteria:

* Primary Ocular Melanoma
* Prior therapy with a Cytotoxic T Lymphocyte Antigen 4 (CTLA-4) or Programmed death- 1 (PD-1) antagonist, or Programmed cell death- ligand 1 (PD-L1) or CD137 agonists
* Symptomatic brain metastases
* History of autoimmune diseases

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2012-11-12 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (32):
- United States (14):
  - Phoenix Children'S Hospital, Phoenix, Arizona
  - Childrens Hospital Of La, Los Angeles, California
  - Children'S Hospital Of Orange County, Orange, California
  - Children'S Hospital Colorado, Aurora, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - James Whitcomb Riley Hospital For Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Of Pittsburgh Medical Center Cancer Center, Pittsburgh, Pennsylvania
  - St. Jude Children'S Research Hospital, Memphis, Tennessee
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
  - Primary Children'S Medical Center, Salt Lake City, Utah
  - University Of Utah, Salt Lake City, Utah
- Local Institution, Ghent, Belgium
- Local Institution, Copenhagen, Denmark
- France (4):
  - Local Institution, Lyon
  - Local Institution, Marseille
  - Local Institution, Nantes
  - Local Institution, Villejuif
- Germany (5):
  - Local Institution, Dortmund
  - Local Institution, Erlangen
  - Local Institution, Hamburg
  - Local Institution, M?nster
  - Local Institution, Münster
- Mexico (3):
  - Local Institution, México, D.F
  - Local Institution, Leon, Guanajato, Guanajuato
  - Local Institution, Df, Mexico City
- Local Institution, Esplugues de Llobregat- Barcelona, Spain
- United Kingdom (3):
  - Local Institution, Bristol, Avon
  - Local Institution, Newcastle, Northumberland
  - Local Institution, Sutton, Surrey

REFERENCES:
- [Derived] Geoerger B, Bergeron C, Gore L, Sender L, Dunkel IJ, Herzog C, Brochez L, Cruz O, Nysom K, Berghorn E, Simsek B, Shen J, Pappo A. Phase II study of ipilimumab in adolescents with unresectable stage III or IV malignant melanoma. Eur J Cancer. 2017 Nov;86:358-363. doi: 10.1016/j.ejca.2017.09.032. Epub 2017 Nov 5. PMID 29100190
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 participants were enrolled in the study. 12 participants received study treatment. 2 participants were enrolled and not treated because they no longer met study criteria.
Groups:
- Ipilimumab 3mg/kg; Ipilimumab 10mg/kg: Ipilimumab was administered intravenously (IV) over 90 minutes on Day 1 of each 21-day cycle for 4 cycles.
Period: Overall Study
Arm/Group | Ipilimumab 3mg/kg | Ipilimumab 10mg/kg
Started | 4 | 8
Completed | 1 | 1
Not Completed | 3 | 7
Not completed — Study drug toxicity | 1 | 5
Not completed — Disease progression | 2 | 2

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab 3mg/kg | Ipilimumab 10mg/kg | Total
Number analyzed (Participants) | 4 | 8 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (1.89) | 14.9 (0.64) | 14.3 (1.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 8 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Rate at 1 Year
Description: Overall Survival (OS) was defined as the time from the start of ipilimumab treatment date to death due to any cause. If a participant had not died, the participant was censored at the time of last contact (last known alive date). OS rates at 1 year were calculated from both Kaplan-Meier estimates and the proportion of participants alive at 1 year following start of treatment.
Time Frame: 1 year following start of treatment (Assessed up to June 2016, approximately 38 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipilimumab 3mg/kg | Ipilimumab 10mg/kg
Number analyzed (Participants) | 4 | 8
percentage of participants
  OS Rate (Kaplan-Meier estimates) | 75.0 [12.8 to 96.1] | 62.5 [22.9 to 86.1]
  OS Rate (Proportion of surviving participants) | 75.0 [19.4 to 99.4] | 62.5 [24.5 to 91.5]

2. Primary Outcome: Percentage of Participants With Severe Immune-Mediated Adverse Reactions (imARs)
Description: The percentage of participants with severe Immune-mediated Adverse Reactions (imARs) was determined by dividing the number of participants with grade 3 or worse imARs by the total number of treated participants and expressing this number as a percentage. imARs were AEs determined by the investigator to have an immune-mediated etiology, including inflammatory events associated with ipilimumab treatment.
Time Frame: From first dose to 90 days after last dose (Assessed up to June 2016, approximately 38 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipilimumab 3mg/kg | Ipilimumab 10mg/kg
Number analyzed (Participants) | 4 | 8
percentage of participants | 25.0 [0.6 to 80.6] | 62.5 [24.5 to 91.5]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate was defined as the percentage of all treated participants with a best overall response of Complete Response (CR), Partial Response (PR), or Stable disease (SD), based on the investigator's assessment per mWHO Criteria.
  CR= Complete disappearance of all non-index lesions. PR= Decrease, relative to baseline, of 50% or greater in the sum of the products of the two largest perpendicular diameters of all index lesions. SD= Does not meet criteria for complete or partial response, in the absence of progressive disease. PD= At least 25% increase in the sum of the products of all index lesions (taking as reference the smallest sum recorded at or following baseline) and/or the appearance of any new lesion(s).
Time Frame: From Day 1 of first subject, first treatment to Day 365 of last subject, first treatment (approximately 36 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab 3mg/kg | Ipilimumab 10mg/kg
Number analyzed (Participants) | 4 | 8
Percentage of participants | 25.0 [0.6 to 80.6] | 37.5 [8.5 to 75.5]

4. Secondary Outcome: Progression Free Survival
Description: Progression-Free Survival was defined as the time from the start of ipilimumab treatment to disease progression or death, whichever occurs first. A participant who died without reported progression was considered to have progressed on their date of death. For participants who remained alive and had not progressed, PFS was censored on the date of the last tumor assessment.
Time Frame: From date of first treatment until disease progression or death (Assessed up to June 2016, approximately 38 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab 3mg/kg | Ipilimumab 10mg/kg
Number analyzed (Participants) | 4 | 8
months | 2.6 [2.3 to 8.5] | 2.9 [0.7 to NA] — Upper 95% CI value was not reached

5. Secondary Outcome: Best Overall Response Rate (BORR)
Description: Best Overall Response Rate (BORR) was defined as the total number of participants with the best overall response of Complete Response (CR) or Partial Response (PR) divided by the total number of treated participants and expressed as a percentage.
  CR= Complete disappearance of all non-index lesions. PR= Decrease, relative to baseline, of 50% or greater in the sum of the products of the two largest perpendicular diameters of all index lesions. SD= Does not meet criteria for complete or partial response, in the absence of progressive disease. PD= At least 25% increase in the sum of the products of all index lesions (taking as reference the smallest sum recorded at or following baseline) and/or the appearance of any new lesion(s).
Time Frame: From Day 1 of first subject, first treatment to Day 365 of last subject, first treatment (approximately 36 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipilimumab 3mg/kg | Ipilimumab 10mg/kg
Number analyzed (Participants) | 4 | 8
percentage of participants | 0.0 [0.0 to 60.2] | 25.0 [3.2 to 65.1]

6. Secondary Outcome: Overall Survival Time
Description: Overall Survival time was defined as the time from the start of ipilimumab treatment date to date of death due to any cause. Participants who had not died were censored at the time of last contact (last known alive date).
Time Frame: From date of first treatment to date of death (Assessed up to June 2016, approximately 38 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab 3mg/kg | Ipilimumab 10mg/kg
Number analyzed (Participants) | 4 | 8
months | 18.2 [8.9 to 18.2] | NA [5.2 to NA] — Median and upper 95% CI values were not reached

ADVERSE EVENTS:
Time Frame: From date of first dose to 90 days after date of last dose, assessed up to study completion (approximately 38 months)
Groups:
- IPILIMUMAB 3 MG/KG; IPILIMUMAB 10 MG/KG: Ipilimumab was administered intravenously (IV) over 90 minutes on Day 1 of each 21-day cycle for 4 cycles.
Arm/Group | IPILIMUMAB 3 MG/KG | IPILIMUMAB 10 MG/KG
Serious Adverse Events (participants affected / at risk) | 1/4 | 6/8
Other Adverse Events (participants affected / at risk) | 4/4 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IPILIMUMAB 3 MG/KG (N=4) | IPILIMUMAB 10 MG/KG (N=8)
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IPILIMUMAB 3 MG/KG (N=4) | IPILIMUMAB 10 MG/KG (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Eyelid pain (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Haematochezia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 6
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 7
Asthenia (General disorders) | 1 | 0
Axillary pain (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 4
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 3
Hepatitis (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Candida nappy rash (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Rotavirus infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Amylase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood albumin decreased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Coagulation factor increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 4
White blood cell count increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 5
Tremor (Nervous system disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.